CLINICAL TRIAL: NCT04174261
Title: Ticagrelor in Remote Ischemic Preconditioning Study
Acronym: TRIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hellenic Society of Interventional Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ESR-14-10310
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Periprocedural Myocardial Infarction
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Intervention Model Description: The TRIP study was a randomized, assessor-blind, active comparator-controlled, clinical trial using a 2×2 factorial design, with 1:1 patient allocation to ticagrelor or clopidogrel and within each treatment a 1:1 allocation to RIPC or control.
Who Masked: Outcomes Assessor
Masking Description: Patient randomization in the ticagrelor and the clopidogrel group took place using sealed, opaque envelopes containing a computer-generated randomization scheme. Using a similar procedure, patients were then randomly assigned to RIPC or no RIPC within 1 hour before the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ticagrelor - Remote Ischemic Preconditioning (Experimental): Ticagrelor 180mg loading dose, and 90mg b.i.d thereafter. 3 cycles of 5-minute ischemia/5-minute reperfusion using a BP cuff around the non-dominant arm
  Interventions: Drug: Ticagrelor; Procedure: Remote Ischemic Preconditioning
- Ticagrelor - Control (Other): Ticagrelor 180mg loading dose, and 90mg b.i.d thereafter. BP-cuff uninflated around the non-dominant arm
  Interventions: Drug: Ticagrelor
- Clopidogrel - Remote Ischemic Preconditioning (Active Comparator): Clopidogel 300mg loading dose, and 75mg q.d. thereafter. 3 cycles of 5-minute ischemia/5-minute reperfusion using a BP cuff around the non-dominant arm
  Interventions: Procedure: Remote Ischemic Preconditioning; Drug: Clopidogrel
- Clopidogrel - Control (Other): Clopidogel 300mg loading dose, and 75mg q.d. thereafter. BP-cuff uninflated around the non-dominant arm
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Preprocedural ticagrelor loading and standard dose thereafter
  Arms: Ticagrelor - Control; Ticagrelor - Remote Ischemic Preconditioning
Procedure: Remote Ischemic Preconditioning — Preprocedural remote ischemic preconditioning on the non-dominant arm
  Arms: Clopidogrel - Remote Ischemic Preconditioning; Ticagrelor - Remote Ischemic Preconditioning
Drug: Clopidogrel — Preprocedural clopidogrel loading and standard dose thereafter
  Arms: Clopidogrel - Control; Clopidogrel - Remote Ischemic Preconditioning

SUMMARY:
Remote ischemic preconditioning (RIPC) reduces periprocedural myocardial injury (PMI) after percutaneous coronary intervention (PCI) through various pathways, including an adenosine-triggered pathway. Ticagrelor inhibits adenosine uptake, thus may potentiate the effects of RIPC.

This randomized trial tested the hypothesis that ticagrelor potentiates the effect of RIPC and reduces PMI, as assessed by post-procedural troponin release

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is often complicated by peri-procedural myocardial injury, with widespread adoption of sensitive cardiac biomarkers assays allowing detection of smaller amounts of myocardial necrosis (1, 2). Peri-procedural cardiac troponin elevation has been associated with new irreversible myocardial injury, detected by delayed-enhancement magnetic resonance imaging (3), and even though the prognostic significance of peri-procedural cardiac troponin elevation has been highly debated (4), several studies have reported that peri-procedural injury is associated with worse prognosis (5, 6).

Peri-procedural myocardial injury attenuation is expected to improve cardiovascular outcomes following PCI, and this could be achieved through such cardioprotective interventions as ischemic preconditioning (IPC) (2). Converging experimental and clinical evidence suggests that the long-established therapeutic potential of remote IPC or ischemic perconditioning may find clinical use in the setting of elective PCI or ST-elevation myocardial infarction (MI)(7-9). Nevertheless, recent clinical trials suggest that the cardioprotective effect of remote IPC is moderate (10, 11), thus demonstrating the need to explore methods to augment it.

The ischemic conditioning signal is considered a summation of signals derived from multiple disparate receptor-ligand interactions, which reaches a threshold once sufficient combined signals are generated (12, 13). Adenosine, with its plasma levels increasing after cellular stresses and ischemia, is a crucial trigger of the preconditioning cascade (14), however it is rapidly taken up by cells through sodium-independent equilibrative nucleoside transporters (ENT 1/2) and sodium-dependent concentrative nucleoside transporters (CNT 2/3) (15).

Experimental data suggest that ticagrelor inhibits cellular reuptake of adenosine, thereby increasing systemic and tissue adenosine levels (15-17). Moreover, the antiplatelet effects of ticagrelor have been shown to be partly mediated by increased extracellular adenosine levels and ticagrelor enhances the hyperemic response to adenosine (16, 18). Clinical evidence suggests that in patients with acute coronary syndromes (ACS) ticagrelor treatment is associated with higher adenosine levels and an augmentation of coronary blood flow velocity in response to adenosine (19, 20). The investigators hypothesized that ticagrelor treatment would potentiate the effects of remote IPC and would thereby reduce peri-procedural myocardial injury and the incidence of post-PCI MI.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Patients (Female and male) ≥ 18 of age
* Patients with NSTE-ACS undergoing coronary angiography, eligible for PCI

Exclusion Criteria:

* Women of childbearing potential
* Severe comorbidity (estimated life expectancy <6 months)
* Baseline cTnI before PCI that is not stable or falling or is > 5 ×99th percentile URL.
* End-stage renal disease(eGFR<15 ml/min/1.73 m2)
* CRUSADE Bleeding Score >50
* Patients with an indication for oral anticoagulation
* On maintenance therapy with ticagrelor or those that have received clopidogrel for less than 3 days
* Use of nicorandil or glibenclamide
* Concomitant theophylline/aminophylline use
* Known contraindications to the use of ticagrelor Hypersensitivity to the active substance or to any of the excipients
* Active pathological bleeding
* History of intracranial haemorrhage
* Moderate to severe hepatic impairment
* Co-administration of ticagrelor with strong CYP3A4 inhibitors (e.g., ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir).
* Patients meeting criteria for immediate or early (<24h) invasive strategy based on the current relevant European Society of Cardiology guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2017-01-29 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
deltaTnI | At the time of PCI / 24 hours post-PCI
  The primary outcome measure of the study was deltaTnI, defined as the difference between cardiac troponin I (cTnI) levels at 24 hours post-PCI and cTnI levels before the procedure.

SECONDARY OUTCOMES:
Peri-procedural MI (type 4a MI) | 24 hours post-PCI
  The prevalence of peri-procedural MI (type 4a MI) according to the third universal definition of MI (5xULN) was a secondary endpoint.
Chest pain during PCI: analog 10-point scale | During the PCI procedure
  Chest pain during PCI was assessed at the post-PCI clinical examination of the subject by an appropriately qualified person, who was unaware of patient's treatment allocation. An analog 10-point scale was used (0: no pain, 10: most severe discomfort ever experienced).
ST-segment deviation during PCI | During the PCI procedure
  ST-segment deviation during PCI was monitored by an appropriately qualified person, who was unaware of patient's treatment allocation. It was defined as the absolute value of ST-segment deviation at 60-80ms after the J-point in mm at the beginning of coronary angiography minus ST-segment deviation at 60-80ms after the J-point in mm during balloon occlusion.

OTHER OUTCOMES:
Bleeding | At the time of PCI / 24 hours post-PCI
  Bleeding, according to the Thrombolysis In Myocardial Infarction (TIMI) criteria, was considered as a safety outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Katsivas, Principal Investigator — Head Cardiology Department, Athens Red Cross Hospital
Locations (1):
- Athens Red Cross Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT04174261/Prot_SAP_000.pdf